CLINICAL TRIAL: NCT03779841
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of Botulinum Toxin Type A (AGN-151607) Injections Into the Epicardial Fat Pads to Prevent Post-Operative Atrial Fibrillation in Patients Undergoing Open-Chest Cardiac Surgery
Brief Title: Botulinum Toxin Type A (AGN-151607) for the Prevention of Post-operative Atrial Fibrillation in Adult Participants Undergoing Open-chest Cardiac Surgery (NOVA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1925-201-008; 2017-004399-68 (EudraCT Number)
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Post-Operative Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- AGN-151607 (250 U) (Experimental): Injections of 50 U were made into each 1 of 5 fat pads. The total injection volume into each fat pad was 1 mL. One-time treatment.
  Interventions: Drug: AGN-151607
- AGN-151607 (125 U) (Experimental): Injections of 25 U were made into each 1 of 5 fat pads. The total injection volume into each fat pad was 1 mL. One-time treatment.
  Interventions: Drug: AGN-151607
- Placebo (Placebo Comparator): Injections of placebo were made into each 1 of 5 fat pads. The total injection volume into each fat pad was 1 mL. One-time treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AGN-151607 — Injections were made into each 1 of 5 fat pads. The total injection volume into each fat pad was 1 mL. One-time treatment.
  Arms: AGN-151607 (125 U); AGN-151607 (250 U)
Drug: Placebo — Injections of placebo were made into each 1 of 5 fat pads. The total injection volume into each fat pad was 1 mL. One-time treatment.
  Arms: Placebo

SUMMARY:
This was a multi-center, randomized, double-blind, placebo-controlled, parallel group, dose-ranging study to evaluate the efficacy and safety of botulinum toxin type A (AGN-151607) injections into the epicardial fat pads, foci of ganglionic plexi, to prevent Post-Operative Atrial Fibrillation (POAF) in patients undergoing open-chest cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form.
* Written informed consent from the participant has been obtained prior to any study-related procedures
* Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable (eg. Written Authorization for Use and Release of Health and Research Study Information [US sites] and written Data Protection consent (European Union sites).
* Participants who are scheduled to undergo open-chest cardiac surgery. Includes: coronary artery bypass graft (CABG) and/or valve repair/replacement. Inclusionary valve repair/replacement procedures for the primary reason for surgery include: Aortic valve repair/replacement, Mitral valve repair/replacement, Combination of aortic and tricuspid valve repair/replacement, Combination of mitral and tricuspid valve repair/replacement CABG/valve combination procedures (when valvular procedure is one of the 4 sub-bulleted procedures immediately above), Left Atrial Appendage (LAA) procedures are allowed if CABG and/or valve repair or replacement is the qualifying surgical procedure, but is not a qualifying surgical procedure on its own.
* A male participant must agree to use contraception until Day 60 and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant (has a negative urine pregnancy result prior to randomization) not breastfeeding, and at least 1 of the following conditions applies: Not a woman of childbearing potential (WOCBP). A WOCBP who agrees to follow the contraceptive guidance until after Day 60.
* In sinus rhythm for the last 48 hours prior to randomization based on standard-of care assessments and study ECGs (note: continuous ECG monitoring for 48 hours is not required; prior history of paroxysmal AF is acceptable)
* Willing to wear an electrocardiogram (ECG) patch for a full 30 days post-surgery and for 7 days after each study visit
* Able, as assessed by the investigator, and willing to follow study instructions and likely to complete required study visit.

Exclusion Criteria:

* Any uncontrolled clinically significant medical condition other than the one under study that, in the investigator's opinion, would put the participant at an unacceptable risk with exposure to botulinum toxin type A.
* Exclusionary valve repair/replacement procedures include: Combination of aortic and mitral valve repair/replacement, Isolated tricuspid valve repair/replacement.
* Any medical condition that may put the participant at increased risk with exposure to botulinum toxin type A, including diagnosed muscular dystrophy (eg, Duchenne's muscular dystrophy), myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, mitochondrial disease, or any other significant disease which might interfere with neuromuscular function.
* Participants with presence or history of any of the following within 3 months prior to the Day 1 visit that may indicate a vulnerable respiratory state per the investigator's clinical judgment: aspiration pneumonia, lower respiratory tract infections, uncontrolled asthma, severe chronic obstructive pulmonary disease, or otherwise compromised respiratory function.
* Permanent/persistent atrial fibrillation (AF)
* Has a known allergy or sensitivity to any botulinum toxin type A preparation. - Has a known allergy or sensitivity to medical adhesive (eg, ECG patch adhesive; hydrogel-based adhesive).
* Severe (> 55 mm left atrial diameter) left atrial enlargement
* Left ventricular ejection fraction (LVEF) < 25%
* Presence or history of symptomatic atrioventricular block > 1st degree within the last 30 days (note: presence of a pacemaker is not exclusionary per se) - Class I or III antiarrhythmic drugs unless proper washout was documented
* Botulinum toxin type A (of any serotype) use within 6 months of randomization
* Has been immunized for any botulinum toxin type A serotype as determined by participant medical history
* Preoperative need for inotropes/vasopressors or intra-aortic balloon pump
* Prior open-chest, sternotomy cardiac surgery - History of ablation for AF
* Planned ablation procedure for AF at the time of surgery
* Emergency surgery
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study
* Participants have diagnostic assessments which in the opinion of the investigator prevent participation in the study
* Impaired prognosis defined as EuroSCORE II > 7% perioperative mortality at screening is exclusionary.
* Females who are pregnant, nursing, or planning a pregnancy during the study
* The participant has a condition or is in a situation which, in the investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (32):
- United States (19):
  - Stanford University School of Med /ID# 236922, Stanford, California
  - Yale New Haven Hospital - Yale School of Medicine /ID# 238221, New Haven, Connecticut
  - Medstar Washington Hospital Center /ID# 234322, Washington D.C., District of Columbia
  - Emory Saint Joseph's Hospital /ID# 234334, Atlanta, Georgia
  - Lutheran Medical Group /ID# 237990, Fort Wayne, Indiana
  - Ochsner Medical Center /ID# 238004, New Orleans, Louisiana
  - University of Maryland Medical Center /ID# 234352, Baltimore, Maryland
  - University of Michigan /ID# 236228, Ann Arbor, Michigan
  - Washington University-School of Medicine /ID# 238121, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center /ID# 237530, Lebanon, New Hampshire
  - Icahn School of Medicine at Mount Sinai - The Mount Sinai Medical Center /ID# 234449, New York, New York
  - Mission Hospital /ID# 237231, Asheville, North Carolina
  - Duke University Medical Center /ID# 234314, Durham, North Carolina
  - East Carolina University /ID# 237820, Greenville, North Carolina
  - Ohio State University Medical Center /ID# 234408, Columbus, Ohio
  - Medical University of South Carolina /ID# 236476, Charleston, South Carolina
  - Baylor Scott & White Research Institute /ID# 235937, Plano, Texas
  - University of Utah /ID# 237601, Salt Lake City, Utah
  - University of Virginia /ID# 237611, Charlottesville, Virginia
- Medizinische Universitaet Wien /ID# 238259, Vienna, Vienna, Austria
- Canada (6):
  - University of Ottawa Heart Institute /ID# 236012, Ottawa, Ontario
  - Toronto General Hospital /ID# 237680, Toronto, Ontario
  - Montreal Heart Insitute /ID# 234859, Montreal, Quebec
  - CHUM - Centre hospitalier de l'Universite de Montréal /ID# 238163, Montreal, Quebec
  - CIUSSS du Nord-de-l'ile-de-Montréal_Hopital du Sacré-Coeur de Montréal /ID# 234316, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université L /ID# 237166, Québec, Quebec
- Asklepios Klinik Harburg-Hamburg /ID# 234855, Hamburg, Germany
- ASST degli Spedali Civili di Brescia /ID# 234861, Brescia, Italy
- Academisch Medisch Centrum /ID# 237113, Amsterdam, Netherlands
- Hospital Clínic. University of Barcelona /ID# 234853, Barcelona, Spain
- Orebro University Hospital Sweden /ID# 236047, Örebro, Örebro County, Sweden
- University Hospital Plymouth NHS Trust /ID# 234423, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Piccini JP, Ahlsson A, Dorian P, Gillinov MA, Kowey PR, Mack MJ, Milano CA, Perrault LP, Steinberg JS, Waldron NH, Adams LM, Bharucha DB, Brin MF, Ferguson WG, Benussi S. Design and Rationale of a Phase 2 Study of NeurOtoxin (Botulinum Toxin Type A) for the PreVention of Post-Operative Atrial Fibrillation - The NOVA Study. Am Heart J. 2022 Mar;245:51-59. doi: 10.1016/j.ahj.2021.10.114. Epub 2021 Oct 20. PMID 34687654

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 323 subjects were randomized, of which 319 received study drug (Safety Population).
Period: Randomized Population
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Started | 108 | 106 | 109
Completed | 105 | 105 | 109
Not Completed | 3 | 1 | 0
Not completed — Did Not Receive Treatment | 3 | 1 | 0
Period: Treated (Safety) Population
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Started | 105 | 105 | 109
Completed | 94 | 87 | 93
Not Completed | 11 | 18 | 16
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 8 | 6
Not completed — Lost to Follow-up | 5 | 9 | 8
Not completed — Death | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U) | Total
Number analyzed (Participants) | 105 | 105 | 109 | 319
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 43 | 42 | 45 | 130
  >=65 years | 62 | 63 | 64 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (6.76) | 66.8 (6.54) | 67.2 (7.01) | 66.9 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 22 | 53
  Male | 91 | 88 | 87 | 266
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 6 | 20
  Not Hispanic or Latino | 99 | 97 | 103 | 299
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 102 | 102 | 105 | 309
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Type of Surgery [Count of Participants; unit: Participants]
  Isolated Coronary Artery Bypass Graft (CABG) Surgery | 65 | 68 | 70 | 203
  Valve only Surgery | 27 | 24 | 27 | 78
  CABG and Valve Surgery | 13 | 13 | 12 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Continuous AF (Atrial Fibrillation or Atrial Flutter) Episode ≥ 30 Seconds During the First 30 Days Post-surgery
Description: At least one episode of continuous AF (atrial fibrillation or atrial flutter) sustained ≥ 30 seconds documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial intensive care unit (ICU) admission date after open-chest cardiac surgery.
Population: All randomized participants who received study treatment and had at least 1 post-dose ECG (by ePatch) by Day 30 post-surgery.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 46.1 | 36.5 | 47.2
Statistical Analysis 1: Comparison: AGN-151607 (125 U); P-values and Risk Ratios (and their corresponding 95% CI) for each pairwise comparison of AGN-151607 versus Placebo are obtained from Cochran-Mantel-Haenszel (CMH) test controlling for type of surgery (presence or absence of valve surgery) and age group (< 65 or ≥ 65 years); Test type: Superiority; p = 0.1612, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.58 to 1.10]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7789, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.79 to 1.37]

2. Secondary Outcome: Percentage of Time Spent in Atrial Fibrillation or Atrial Flutter (AF Burden) During the First 30 Days Post-surgery
Description: The proportion of time an individual is in AF (atrial fibrillation or atrial flutter) during a monitoring period (expressed as a percentage) calculated as (the total time spent in AF during the first 30 days post-surgery divided by the total time of analyzable data obtained from the ECG patch during the first 30 days post-surgery) multiplied by 100. The calculation excludes continuous AF episodes < 30 seconds in duration.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of time | 4.84 (14.898) | 4.41 (14.976) | 5.45 (15.821)
Statistical Analysis 1: Comparison: AGN-151607 (125 U); P-value is obtained from stratified Wilcoxon (Van Elteren) test versus Placebo with type of surgery (presence or absence of valve surgery) and age group (< 65 or ≥ 65 years) as stratification factors; Test type: Superiority; p = 0.2972, stratified Wilcoxon (Van Elteren)
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8722, stratified Wilcoxon (Van Elteren)

3. Secondary Outcome: Percentage of Participants With at Least 1 Event of Symptomatic AF (Atrial Fibrillation or Atrial Flutter) During the First 30 Days Post-surgery
Description: At least 1 event of symptomatic AF (atrial fibrillation or atrial flutter) (symptoms occurring within 2 hours of an AF episode). For symptomatic AF, symptoms that occur in the interval that starts two hours prior to the onset of the AF episode and ends two hours after the conclusion of the AF episode will meet the definition of "within 2 hours of an AF episode".
  AF episode ≥ 30 seconds.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 13.7 | 13.5 | 13.2
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9814, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.50 to 1.96]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9715, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.50 to 1.97]

4. Secondary Outcome: Time to First Occurrence of AF (Atrial Fibrillation or Atrial Flutter) During the First 30 Days Post-surgery
Description: Amount of time (days) to first AF (atrial fibrillation or atrial flutter) occurrence defined by first episode of AF lasting for ≥ 30 seconds.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
Days | NA [9.1 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [13.2 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: AGN-151607 (125 U); P-value is from stratified log-rank test versus Placebo with type of surgery (presence or absence of valve surgery) and age group (< 65 or ≥ 65 years) as stratification factors; Test type: Superiority; p = 0.1281, Log Rank
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.8820, Log Rank

5. Secondary Outcome: Percentage of Participants With at Least 1 Continuous AF (Atrial Fibrillation or Atrial Flutter) Episode ≥ 2 Minutes During the First 30 Days Post-surgery
Description: At least one episode of continuous AF (atrial fibrillation or atrial flutter) sustained ≥ 2 minutes documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 45.1 | 35.6 | 46.2
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1623, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.57 to 1.10]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7776, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.78 to 1.39]

6. Secondary Outcome: Percentage of Participants With at Least 1 Continuous AF (Atrial Fibrillation or Atrial Flutter) Episode ≥ 5 Minutes During the First 30 Days Post-surgery
Description: At least one episode of continuous AF (atrial fibrillation or atrial flutter) sustained ≥ 5 minutes documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 44.1 | 34.6 | 46.2
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1603, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.56 to 1.10]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6706, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.06, 95% CI 2-sided [0.80 to 1.42]

7. Secondary Outcome: Percentage of Participants With at Least 1 Continuous AF (Atrial Fibrillation or Atrial Flutter) Episode ≥ 6 Minutes During the First 30 Days Post-surgery
Description: At least one episode of continuous AF (atrial fibrillation or atrial flutter) sustained ≥ 6 minutes documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 43.1 | 33.7 | 45.3
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1583, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.55 to 1.10]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6694, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.80 to 1.43]

8. Secondary Outcome: Percentage of Participants With at Least 1 Continuous AF (Atrial Fibrillation or Atrial Flutter) Episode ≥ 30 Minutes During the First 30 Days Post-surgery
Description: At least one episode of continuous AF (atrial fibrillation or atrial flutter) sustained ≥ 30 minutes documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 38.2 | 30.8 | 39.6
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2578, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.55 to 1.18]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7526, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.76 to 1.47]

9. Secondary Outcome: Percentage of Participants With at Least 1 Continuous AF (Atrial Fibrillation or Atrial Flutter) Episode ≥ 1 Hour During the First 30 Days Post-surgery
Description: At least one episode of continuous AF (atrial fibrillation or atrial flutter) sustained ≥ 1 hour documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 37.3 | 29.8 | 37.7
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2549, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.55 to 1.18]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8544, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.73 to 1.45]

10. Secondary Outcome: Percentage of Participants With at Least 1 Continuous AF (Atrial Fibrillation or Atrial Flutter) Episode ≥ 4 Hours During the First 30 Days Post-surgery
Description: At least one episode of continuous AF (atrial fibrillation or atrial flutter) sustained ≥ 4 hours documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 32.4 | 24.0 | 26.4
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1718, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.74, 95% CI 2-sided [0.48 to 1.14]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3801, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.54 to 1.27]

11. Secondary Outcome: Percentage of Participants With at Least 1 Continuous AF (Atrial Fibrillation or Atrial Flutter) Episode ≥ 6 Hours During the First 30 Days Post-surgery
Description: At least one episode of continuous AF (atrial fibrillation or atrial flutter) sustained ≥ 6 hours documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 25.5 | 22.1 | 20.8
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5531, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.54 to 1.39]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4213, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.51 to 1.33]

12. Secondary Outcome: Percentage of Participants With at Least 1 Continuous AF (Atrial Fibrillation or Atrial Flutter) Episode ≥ 12 Hours During the First 30 Days Post-surgery
Description: At least one episode of continuous AF (atrial fibrillation or atrial flutter) sustained ≥ 12 hours documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 15.7 | 14.4 | 17.0
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8040, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.49 to 1.73]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7573, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.61 to 1.98]

13. Secondary Outcome: Percentage of Participants With at Least 1 Continuous AF (Atrial Fibrillation or Atrial Flutter) Episode ≥ 24 Hours During the First 30 Days Post-surgery
Description: At least one episode of continuous AF (atrial fibrillation or atrial flutter) sustained ≥ 24 hours documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 9.8 | 6.7 | 12.3
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4065, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.69, 95% CI 2-sided [0.28 to 1.67]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5257, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.28, 95% CI 2-sided [0.60 to 2.70]

14. Secondary Outcome: Percentage of Participants With at Least 1 Continuous Atrial Fibrillation (Excluding Atrial Flutter) Episode ≥ 30 Seconds During the First 30 Days Post-surgery
Description: At least one episode of continuous atrial fibrillation (excluding atrial flutter) sustained ≥ 30 seconds documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 43.1 | 33.7 | 42.5
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1612, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.55 to 1.11]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9966, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.74 to 1.35]

15. Secondary Outcome: Percentage of Participants With at Least 1 Continuous Atrial Flutter Episode ≥ 30 Seconds During the First 30 Days Post-surgery
Description: At least one episode of continuous atrial flutter sustained ≥ 30 seconds documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 12.7 | 8.7 | 15.1
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3374, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.68, 95% CI 2-sided [0.30 to 1.52]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5403, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.23, 95% CI 2-sided [0.62 to 2.45]

16. Secondary Outcome: Percentage of Participants With at Least 1 Continuous Atrial Tachycardia Episode (Defined as the Duration of the Longest Supraventricular Tachycardia [SVT] Run) ≥ 30 Seconds During the First 30 Days Post-surgery
Description: At least one episode of continuous atrial tachycardia sustained ≥ 30 seconds documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 2.9 | 11.5 | 7.5
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0163, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 3.94, 95% CI 2-sided [1.16 to 13.42]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1101, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 2.70, 95% CI 2-sided [0.76 to 9.64]

17. Secondary Outcome: Percentage of Participants With at Least 1 Continuous Episode of Either Atrial Fibrillation or Atrial Flutter or Atrial Tachycardia ≥ 30 Seconds During the First 30 Days Post-surgery
Description: At least one episode of continuous atrial fibrillation or atrial flutter or atrial tachycardia sustained ≥ 30 seconds documented by monitoring ECG measurements using ECG patches (ePatch) placed on the participant's chest.
Time Frame: First 30 days following the initial ICU admission date after open-chest cardiac surgery.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
Number analyzed (Participants) | 102 | 104 | 106
percentage of participants | 48.0 | 41.3 | 51.9
Statistical Analysis 1: Comparison: AGN-151607 (125 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3339, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.64 to 1.16]
Statistical Analysis 2: Comparison: AGN-151607 (250 U); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4614, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.85 to 1.42]

ADVERSE EVENTS:
Time Frame: The length of this study was up to 367 days post single dose study treatment, plus up to 28 days before the first study day (randomization, Day 1). Of the 323 subjects enrolled and included in the All-Cause Mortality table, 4 did not receive treatment and, therefore, did not go beyond the 28-Day screening period. The median time followed for the 319 subjects who received a single treatment of Placebo, AGN-151607 125 Units, or AGN-151607 250 Units was 371.0, 372.0 and 371.0 days, respectively.
Arm/Group | Placebo | AGN-151607 (125 U) | AGN-151607 (250 U)
All-Cause Mortality (participants affected / at risk) | 1/108 | 0/106 | 2/109
Serious Adverse Events (participants affected / at risk) | 36/105 | 38/105 | 28/109
Other Adverse Events (participants affected / at risk) | 86/105 | 84/105 | 94/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=105) | AGN-151607 (125 U) (N=105) | AGN-151607 (250 U) (N=109)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
BLOOD LOSS ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
COAGULOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 6 (7) | 6 (6) | 4 (6)
ATRIAL FLUTTER (Cardiac disorders) | 5 (5) | 1 (1) | 5 (5)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY PERFORATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
NODAL RHYTHM (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
DIPLOPIA (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
AORTO-OESOPHAGEAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 2 (2) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
COLONIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
MEDIASTINITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CORONARY SINUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PERIPROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TRANSFUSION-RELATED ACUTE LUNG INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
VASCULAR PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
ELECTROENCEPHALOGRAM ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
BELL'S PALSY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
FACIAL PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MYASTHENIA GRAVIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 3 (3) | 1 (2)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (3) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIAPHRAGMATIC PARALYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 2 (2)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC PERFORATION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=105) | AGN-151607 (125 U) (N=105) | AGN-151607 (250 U) (N=109)
ANAEMIA (Blood and lymphatic system disorders) | 27 (28) | 19 (20) | 30 (30)
ATRIAL FIBRILLATION (Cardiac disorders) | 32 (38) | 31 (37) | 35 (40)
ATRIAL FLUTTER (Cardiac disorders) | 6 (6) | 5 (6) | 7 (7)
BRADYCARDIA (Cardiac disorders) | 4 (4) | 7 (8) | 4 (4)
PALPITATIONS (Cardiac disorders) | 7 (10) | 4 (6) | 6 (6)
SINUS TACHYCARDIA (Cardiac disorders) | 7 (8) | 1 (1) | 2 (2)
TACHYCARDIA (Cardiac disorders) | 4 (4) | 4 (6) | 12 (12)
CONSTIPATION (Gastrointestinal disorders) | 10 (10) | 7 (9) | 6 (6)
NAUSEA (Gastrointestinal disorders) | 25 (25) | 25 (27) | 29 (30)
VOMITING (Gastrointestinal disorders) | 4 (4) | 2 (2) | 7 (7)
FATIGUE (General disorders) | 7 (8) | 3 (3) | 5 (5)
OEDEMA PERIPHERAL (General disorders) | 13 (15) | 10 (11) | 10 (10)
PYREXIA (General disorders) | 2 (2) | 8 (8) | 5 (6)
COVID-19 (Infections and infestations) | 5 (5) | 10 (12) | 6 (6)
URINARY TRACT INFECTION (Infections and infestations) | 4 (4) | 6 (7) | 6 (6)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 20 (20) | 20 (21) | 21 (21)
VASOPLEGIA SYNDROME (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 13 (13)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 14 (16) | 17 (19) | 17 (17)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 18 (19) | 24 (24) | 23 (23)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 9 (9)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 5 (5) | 6 (6) | 7 (7)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 12 (12) | 11 (12) | 9 (9)
DIZZINESS (Nervous system disorders) | 8 (10) | 4 (4) | 5 (5)
ANXIETY (Psychiatric disorders) | 6 (6) | 3 (4) | 5 (5)
DELIRIUM (Psychiatric disorders) | 2 (2) | 2 (2) | 6 (6)
INSOMNIA (Psychiatric disorders) | 16 (16) | 17 (17) | 12 (12)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 11 (11) | 18 (20)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3) | 7 (7)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 3 (4) | 13 (13)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 10 (11) | 22 (24)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 6 (6)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 6 (6)
HYPERTENSION (Vascular disorders) | 8 (9) | 7 (7) | 6 (6)
HYPOTENSION (Vascular disorders) | 15 (18) | 10 (10) | 17 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT03779841/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT03779841/SAP_001.pdf